CLINICAL TRIAL: NCT05297331
Title: A Prospective Assessment of the Perioperative Parameter and Treatment Outcomes of Urinary Calculi - International Registry
Brief Title: Renal Stone Treatment Global Registry
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2021.684
Record Dates: First submitted 2022-03-09; First posted 2022-03-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; ESWL; RIRS; flexible ureteroscopy; PCNL; FANS; flexible and navigable suction ureteral access sheath; intrarenal pressure; IRP; intrarenal temperature; IRT
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- FLEXOR-FANS (flexible and navigable suction ureteral access sheath): Cohort of flexible ureteroscopy with flexible and navigable suction ureteral access sheath (fURS FANS) will be studied
- DISS (Direct in scope suction): Cohort of flexible ureteroscopy with direct in scope suction (DISS) will be studied
- Flexible ureteroscopy - IRP / IRT: Cohort of flexible ureteroscopy with and without real-time intrarenal pressure (IRP) monitoring and/or intrarenal temperature (IRT) will be studied
- Shockwave lithotripsy (SWL): Cohort of extracorporeal shockwave lithotripsy (SWL) will be studied
- Percutaneous nephrolithotomy (PCNL): Cohort of percutaneous nephrolithotomy with or without intrarenal pressure and temperature monitoring will be studied.

SUMMARY:
This is an international prospective data registry to assess the treatment outcomes and complications of different treatment approaches for different surgical treatment of urolithiasis.

DETAILED DESCRIPTION:
Renal stone is a common condition, and many patients suffered from recurrent diseases and required multiple interventions in their lifetime. Currently, there are many treatment options available for stone treatment, including shockwave lithotripsy, ureteroscopy, percutaneous nephrolithotomy etc.

Different treatment approaches will result in different treatment successful rate and also potential adverse effects to patients. The main challenge for stone management is the decision on the best treatment approach for individual stone of each patient. This is because for the same type of stone (such as lower caliceal stone or upper ureteric stone), different surgical treatment could be applied. The decision will depend on various patients (such as age, premorbid etc.) and stone factors (such as size, density etc) and also patients' preference.

New advances in technology have improved treatment outcomes for urolithiasis, such as single use flexible ureteroscopes, flexible and navigable ureteral access sheaths (FANS), direct in scope suction (DISS), intrarenal pressure (IRP) and intrarenal temperature (IRT) monitoring devices, new lasers and pulse modulation, etc.

Therefore, in order to have more information to guide treatment decision during discussion with patients, a prospective data registry is created to assess the treatment outcomes and complications of different treatment approaches in our hospital clusters. This information will be important for audit, treatment comparison and also patient education.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the age of 18 or above

Exclusion Criteria:

* Patient is unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with urinary stones and planned for surgery (including shockwave lithotripsy, ureteroscopy, percutaneous nephrolithotomy (PCNL), laparoscopic ureterolithiasis, open stone procedures etc) in the hospitals will be identified and then enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Target Stone status | postoperative, at 1 and/or 3 months
  stone free rate

SECONDARY OUTCOMES:
Intraoperative parameters | intraoperative
  Including irrigation and suction and laser settings and devices, laser consumption and efficacy, fluoroscopy dosage and time, equipment (ureteral access sheath size and lengths, ureteroscopy sizes, stone basket) utilised; exit strategy; intraoperative complications if noted; ergonomics
Treatment related complication | Thirty days after the operation
  The 30-day complications will be graded according to the Clavien-Dindo classification
Recurrence of stone | At 12 months
  Stone recurrence rate
QOL and pain scores | preoperative, postoperative on day 0 and at follow up
  Pain VAS scores and QOL assessment

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
  - North District Hospital, Sheung Shui

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gauhar V, Traxer O, Fong KY, Sietz C, Chew BH, Bin Hamri S, Gokce MI, Gadzhiev N, Yuen SKK, Malkhasyan V, Ragoori D, Tanidir Y, Somani BK, Castellani D. Comparing Thulium Fiber Versus High-Power Holmium Laser Lithotripsy Combined with the Flexible and Navigable Suction Access Sheath in Flexible Ureteroscopy for Kidney Stone Disease: A Propensity Score Matched Analysis by the Global FANS Collaborative Group. J Endourol. 2025 Jan;39(1):42-49. doi: 10.1089/end.2024.0653. Epub 2024 Dec 16. PMID 39676748
- [Background] Yuen SKK, Zhong W, Chan YS, Castellani D, Bhojani N, Agarwal MS, Tokas T, Croghan S, Jung H, Herrmann T, Somani B, Gauhar V; Global Research on Intra-renal Pressure Collaborative Group. Current utility, instruments, and future directions for intra-renal pressure management during ureteroscopy: scoping review by global research in intra-renal pressure collaborative group initiative. Ther Adv Urol. 2025 Jan 31;17:17562872251314809. doi: 10.1177/17562872251314809. eCollection 2025 Jan-Dec. PMID 39896048
- [Background] Zhu W, Yuen SKK, Cao J, et al. Intrarenal pressure monitoring via flexible and navigable suction ureteral access sheath in retrograde intrarenal surgery: A preclinical animal study and a pilot clinical study. Clinical and Translational Discovery. 2025;5:e70031doi:10.1002/ctd2.70031
- [Background] Nedbal C, Yuen SKK, Akram M, Keller EX, Martinez BB, Philip J, Emiliani E, Li JKM, Stracci D, Gauhar V, Castellani D, Somani BK. First clinical evaluation of a flexible digital ureteroscope with direct in scope suctioning system (Pusen DISS 7.5Ch): prospective multicentric feasibility study. World J Urol. 2024 Oct 3;42(1):560. doi: 10.1007/s00345-024-05275-9. PMID 39361036
- [Background] Gauhar V, Traxer O, Castellani D, Sietz C, Chew BH, Fong KY, Hamri SB, Gokce MI, Gadzhiev N, Galosi AB, Yuen SKK, El Hajj A, Ko R, Zawadzki M, Sridharan V, Lakmichi MA, Corrales M, Malkhasyan V, Ragoori D, Soebhali B, Tan K, Chai CA, Tursunkulov AN, Tanidir Y, Persaud S, Elshazly M, Kamal W, Tefik T, Shrestha A, Tiong HC, Somani BK. Could Use of a Flexible and Navigable Suction Ureteral Access Sheath Be a Potential Game-changer in Retrograde Intrarenal Surgery? Outcomes at 30 Days from a Large, Prospective, Multicenter, Real-world Study by the European Association of Urology Urolithiasis Section. Eur Urol Focus. 2024 Dec;10(6):975-982. doi: 10.1016/j.euf.2024.05.010. Epub 2024 May 24. PMID 38789313
- [Background] Yuen SKK, Traxer O, Wroclawski ML, Gadzhiev N, Chai CA, Lim EJ, Giulioni C, De Stefano V, Nedbal C, Maggi M, Sarica K, Castellani D, Somani B, Gauhar V. Scoping Review of Experimental and Clinical Evidence and Its Influence on Development of the Suction Ureteral Access Sheath. Diagnostics (Basel). 2024 May 16;14(10):1034. doi: 10.3390/diagnostics14101034. PMID 38786332
- [Background] Talyshinskii A, Tzelves L, Ventimiglia E, Yuen SKK, Gauhar V, Traxer O, Somani B. Technological innovation and revolution with single-use digital flexible ureteroscopes: a review from section of EAU Endourology. Curr Opin Urol. 2025 Jul 1;35(4):360-367. doi: 10.1097/MOU.0000000000001260. Epub 2025 Jan 7. PMID 39774241
- [Background] Gauhar V, Somani BK, Seitz C, Castellani D, Tefik T, Persaud S, Ragoori D, Gauhar V, Tan K, Lakmichi MA, Gadzhiev N, Malkhasyan V, Kamal W, Tanidir Y, Chai CA, Tursunkulov AN, Farahat Y, Keller EX, Chew BH, Herrmann T, Traxer O, Yuen SKK. A Global Survey to Assess Urologists' Attitudes Towards Suction Technology in Endourology by the European Association of Urology Section of Endourology and Progressive Endourological Association for Research and Leading Solutions. Urology. 2025 Mar;197:42-50. doi: 10.1016/j.urology.2024.12.009. Epub 2024 Dec 16. PMID 39674378
- [Background] Chan SW, Ng CF, Man CW, Chung R, Li SK. A report on a randomly sampled questionnaire survey about renal stone disease in Hong Kong. Hong Kong Med J. 2008 Dec;14(6):427-31. PMID 19060340
- [Background] Taguchi K, Cho SY, Ng AC, Usawachintachit M, Tan YK, Deng YL, Shen CH, Gyawali P, Alenezi H, Basiri A, Bou S, Djojodemedjo T, Sarica K, Shi L, Singam P, Singh SK, Yasui T. The Urological Association of Asia clinical guideline for urinary stone disease. Int J Urol. 2019 Jul;26(7):688-709. doi: 10.1111/iju.13957. Epub 2019 Apr 24. PMID 31016804
- [Background] Li JK, Teoh JY, Ng CF. Updates in endourological management of urolithiasis. Int J Urol. 2019 Feb;26(2):172-183. doi: 10.1111/iju.13885. Epub 2018 Dec 21. PMID 30575154
- [Background] Ng CF. The effect of age on outcomes in patients undergoing treatment for renal stones. Curr Opin Urol. 2009 Mar;19(2):211-4. doi: 10.1097/mou.0b013e32831e16b7. PMID 19195134
- [Background] Anagnostou T, Thompson T, Ng CF, Moussa S, Smith G, Tolley DA. Safety and outcome of percutaneous nephrolithotomy in the elderly: retrospective comparison to a younger patient group. J Endourol. 2008 Sep;22(9):2139-45. doi: 10.1089/end.2007.0432. PMID 18811570
- [Background] Ng CF, Wong A, Tolley DA. A single-center experience of the usefulness of caliceal-pelvic height in three different lithotripters. J Endourol. 2008 Jul;22(7):1409-15. doi: 10.1089/end.2006.0448. PMID 18690807
- [Background] Ng CF, Luke S, Chiu PK, Teoh JY, Wong KT, Hou SS. The effect of renal cortical thickness on the treatment outcomes of kidney stones treated with shockwave lithotripsy. Korean J Urol. 2015 May;56(5):379-85. doi: 10.4111/kju.2015.56.5.379. Epub 2015 Apr 28. PMID 25964839